CLINICAL TRIAL: NCT01136642
Title: Assessing Top Down and Bottom Up Attention Mechanisms in Smokers Using Nicotine Nasal Spray
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Purpose: Other
Other Study IDs: 999910459; 10-DA-N459
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2012-11-13

CONDITIONS: Drug Addiction; Nicotine Dependence
Keywords: Nicotine; Nicotine Nasal Spray; Attention; Smoking
MeSH Terms: conditions — Substance-Related Disorders; Tobacco Use Disorder; Smoking | interventions — Nicotine

INTERVENTIONS:
Drug: Nicotrol

SUMMARY:
Background:

* Smoking is the leading cause of preventable death in the United States, and researchers are interested in gaining a better understanding of the perceived beneficial effects of nicotine to help improve treatment strategies for nicotine dependence. Understanding the conditions under which nicotine improves attention and cognitive processing may provide more useful information for this research.
* The ability to pay attention and filter relevant from irrelevant stimuli is central to all aspects of information-processing. Top-down and bottom-up attentional processes illustrate how the brain combines stimuli and goal-directed behaviors. Bottom-up processing is an unconscious response to sensory input; for instance, when the eyes automatically focus on a prominent image in a picture. Top-down processing is a conscious response to drive attention toward specific stimuli; for instance, when a person is asked to focus on a less immediately noticeable image in a picture. Researchers are interested in determining whether nicotine improves cognitive performance by acting on top-down or bottom-up attentional mechanisms.

Objectives:

- To investigate the effect of nicotine on the top-down and bottom-up mechanisms of attention in cigarette smokers.

Eligibility:

- Current smokers (at least 10 cigarettes per day for at least 1 year) between 18 and 55 years of age.

Design:

* This study will involve one training session and four experimental sessions.
* During the training session, participants will receive a sample dose of the nicotine nasal spray used in the study to determine if they can tolerate the effects.
* For each experimental session, participants will receive one dose of nicotine nasal spray (1 mg, 2 mg, or 3 mg) or placebo spray, followed by blood pressure and heart rate monitoring, performance of an attentional test, and questionnaires to rate participants perception of nicotine effectiveness. Participants may receive different doses at different sessions, and will not be told which dose they will receive at any given point.

DETAILED DESCRIPTION:
Objective:

The objective is to investigate the dose-response effect of nicotine on the top-down and bottom-up mechanisms of attention in cigarette smokers.

Study population:

Male and nonpregnant-female smokers 18 to 55 years of age.

Design:

This study is a double-blind, placebo controlled trial of nicotine or placebo nasal sprays. Participants have five visits: a training session and four experimental sessions. Each participant receives a test dose of the nasal spray immediately following the training session to ascertain tolerability and become familiarized with the effect of the spray. One dose (0, 1.0, 2.0 or 3.0 mg) of nicotine nasal spray is administered at the beginning of each experimental session followed by the test battery.

Outcome Measures:

Outcome measures are vital signs, ratings of mood and drug effect, and performance (accuracy, response time) on a test of selective attention.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. 18-55 year old male and female cigarette smokers
  2. smoke a minimum of 10 cigarettes per day for at least 1 year

     --Drug Use Survey
  3. estimated IQ score greater than or equal to 85

     --Weschsler Abbreviated Scale of Intelligence (WASI; raw vocabulary cutoff 49)
  4. urine cotinine concentration greater than or equal 100 ng/ml

     * NicAlert reading greater than or equal to 3

EXCLUSION CRITERIA:

1. definite plan to quit smoking in next 30 days
2. consumption of more than 15 alcoholic drinks per week during the past month
3. use of any illicit drugs more than twice per week during the past month

   --Drug Use Survey (items 2-4)
4. pregnant or nursing

   --Urine pregnancy test
5. HIV positive

   --Oral HIV test
6. untreated cardiovascular or pulmonary disease
7. use of nicotine replacement products, bupropion or varenicline, in the past 3 months if specifically used to stop smoking
8. Past history of schizophrenia or bipolar disorder.

   Current Major Depression Disorder, Diagnosis or treatment for Major Depressive Disorder in past 12 months. (H&P)

   Evidence of current ADHD by current diagnosis or medication or score on Adult Symptom Rating Scale; (> 16 on pt A or B must be evaluated by a counselor)
   * SCL-90 > 65 (must be evaluated by a counselor)
   * Beck Depression Inventory-II score greater than or equal to 14 (must be evaluated by a counselor)
9. vital signs (must be outside these parameters on more than two occasions separated by at least one day):

   * systolic blood pressure: minimum 95, maximum 160 mm Hg
   * diastolic blood pressure: minimum 40, maximum 95 mm Hg
   * pulse: minimum 50, maximum 105 bpm
   * respirations: minimum 8, maximum 24 breaths per minute
10. nasal passages: no pathology that would preclude administration of nasal spray
11. under the influence of a drug or alcohol at experimental sessions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2010-01-21; Study Completion 2012-11-13 (Actual)

PRIMARY OUTCOMES:
Performance (accuracy response time) on a test of selective attention.

SECONDARY OUTCOMES:
Vital signs, ratings of mood and drug effect.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Myers, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States